CLINICAL TRIAL: NCT00542893
Title: A Randomized, Open-label, Cross-over Pharmacokinetic Study of Dacarbazine in Combination With Genasense® in Subjects With Advanced Melanoma
Brief Title: A Phase I, Randomized, Open-label, Cross-over, Pharmacokinetic Study of Genasense With and Without Dacarbazine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genta Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GPK105
Record Dates: First submitted 2007-10-10; First posted 2007-10-12 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Advanced Melanoma
Keywords: bcl-2; CFR; DTIC; ECOG; EMEA; MedDRA; NCI CTC; SAE
MeSH Terms: interventions — oblimersen; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Cycle 1: DTIC 1000 mg/m2 Cycle 2: Genasense 7 mg/kg/day for 5 days followed by DTIC 1000 mg/m2
  Interventions: Drug: Genasense® (G3139, oblimersen sodium); Drug: DTIC alone; then Genasense followed by DTIC
- Group 2 (Experimental): Cycle 1: Genasense 7 mg/kg/day for 5 days followed by DTIC 1000 mg/m2 Cycle 2: DTIC 1000 mg/m2
  Interventions: Drug: Genasense® (G3139, oblimersen sodium); Drug: Genasense followed by DTIC; then DTIC alone

INTERVENTIONS:
Drug: Genasense® (G3139, oblimersen sodium)
Drug: Genasense followed by DTIC; then DTIC alone — Cycle 1: Genasense 7 mg/kg/day for 5 days followed by DTIC 1000 mg/m2 Cycle 2: DTIC 1000 mg/m2
  Arms: Group 2
Drug: DTIC alone; then Genasense followed by DTIC — Cycle 1: DTIC 1000 mg/m2 Cycle 2: Genasense 7 mg/kg/day for 5 days followed by DTIC 1000 mg/m2
  Arms: Group 1

SUMMARY:
This clinical drug-drug interaction study is being conducted to evaluate the pharmacokinetics of dacarbazine(DTIC) when administered in combination with Genasense

ELIGIBILITY:
Inclusion Criteria:

* Metastatic Stage IV disease, or Stage III disease that is not surgically resectable
* ECOG Performance Status of 0, 1, or 2
* Life expectancy of at least 12 weeks
* Adequate venous access
* Agreement to practice effective method of birth control

Exclusion Criteria:

* Less than 3 weeks of recovery from prior major surgery or other therapy, including radiation therapy, chemotherapy, or immunotherapy, or cytokine, biologic, or vaccine therapy
* Significant medical disease
* Known hypersensitivity to phosphorothioate-containing oligonucleotides
* Known hypersensitivity to DTIC
* Pregnancy/Lactation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2006-04; Study Completion 2007-09 (Actual)